CLINICAL TRIAL: NCT02077946
Title: A Retrospective Database Assessment of Clinical Effectiveness in Type 2 Diabetes Patients Treated With Liraglutide From Primary Care Centers in Sweden
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-4161; U1111-1151-9632 (Other: WHO)
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Sitagliptin Phosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liraglutide / Sitagliptin
  Interventions: Drug: liraglutide; Drug: sitagliptin

INTERVENTIONS:
Drug: liraglutide — No treatment given.
Drug: sitagliptin — No treatment given.

SUMMARY:
This trial is conducted in Europe. The aim of this study is to investigate a retrospective database assessment of clinical effectiveness in type 2 diabetes patients treated with liraglutide from primary care centers in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Patients from EMR (electronic medical record) system in the primary care in Sweden
* Patients equal to or more than 18 years of age
* Starting treatment with liraglutide or sitagliptin from January 2010 to December 2013
* Minimum of 180 days of prior follow-up/history within the database before their index date

Exclusion Criteria:

* Patients with cancer, end stage liver disease, end stage renal failure (non-diabetes related)
* Female patients with gestational diabetes during pregnancy
* Patients with previous GLP-1 (glucagon-like peptide-1) or DPP-IV (dipeptidyl peptidase-4 ) inhibitor use, i.e. patients should be incretin naïve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be analyzed for patients with type 2 diabetes treated with liraglutide or sitagliptin from January 2010 to December 2013, with a treatment length of 180 days.
Sampling Method: Non-Probability Sample
Enrollment: 1059 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2014-09-03 (Actual); Study Completion 2014-09-03 (Actual)

PRIMARY OUTCOMES:
Percent (%) of patients achieving at least 1 %-point HbA1c (glycosylated haemoglobin) reduction | Day 0, Day 180

SECONDARY OUTCOMES:
Percent (%) of patients with HbA1c (glycosylated haemoglobin) reduction at least 1 %-point and weight reduction at least 3% (NICE clinical guidelines, liraglutide only) | Day 0, Day 180
HbA1c (NGSP standard, in %) change | Day 0, Day 180
Change in weight (in kilograms) | Day 0, Day 180
Change in blood pressure (systolic, in mmHg) | From baseline to 180 days of therapy
Change in lipids (HDL, LDL and triglycerides, in mmol/L) | Day 0, Day 180
Change in creatinine | Day 0, Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Malmo, Sweden

REFERENCES:
- [Background] Lind M, Matsson PO, Linder R, Svenningsson I, Jorgensen L, Ploug UJ, Gydesen H, Dorkhan M, Larsen S, Johansson G. Clinical Effectiveness of Liraglutide vs Sitagliptin on Glycemic Control and Body Weight in Patients with Type 2 Diabetes: A Retrospective Assessment in Sweden. Diabetes Ther. 2016 Jun;7(2):321-33. doi: 10.1007/s13300-016-0173-z. Epub 2016 May 23. PMID 27216947
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com